CLINICAL TRIAL: NCT04259359
Title: Predominant Sensitizations to Single Bee Venom Allergens as a Risk Factor for Therapy Failure
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 31-238 ex 18/19 (PREDICT)
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Bee Venom Allergy
MeSH Terms: conditions — Venom Hypersensitivity | interventions — Arthropod Venoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who will be treated with bee venom immunotherapy
  Interventions: Drug: Insect Venom

INTERVENTIONS:
Drug: Insect Venom — Patients will be treated with bee venom immunotherapy (protocol can be selected by patient). Blood samples are taken before starting VIT to determine specific immunoglobulin E (sIgE) Levels for bee venom components. Patients are sting challenged and the outcome will be recorded.

SUMMARY:
Venom immunotherapy (VIT) is an established treatment for Hymenoptera venom allergy and provides long-term protection from further generalized reactions in almost all patients. However, it is still unclear why bee VIT is less effective than vespid VIT.

The preliminary data show that not only predominant Api m 10 sensitization but also other predominant sensitizations may be relevant as risk factors for treatment failure. Interestingly, all patients with a predominant Api m 10 sensitization who received bee VIT with a venom preparation with a supposed lack of Api m 10 tolerated sting challenges. Therefore, a multicenter study with a sufficient number of patients with treatment failure is urgently required, to clarify if predominant sensitization to a bee venom allergen is a risk factor for treatment failure.

If predominant sensitization is a risk factor and caused by underrepresented components in bee venom preparations used for VIT, bee venom preparations may be optimized in the future and patients would benefit from a more effective VIT.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent male and female subjects aged from 18 to 70 years with a history of a systemic anaphylactic sting reaction (≥ grade I according to the classification of Ring and Messmer) after bee stings, who will receive bee venom immunotherapy

Exclusion Criteria:

* Contraindications to VIT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be treated with bee venom immunotherapy
Sampling Method: Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate whether predominant sensitization to Api m 10 is a risk factor for treatment failure. | depends on the protocol used for VIT and the date of the sting challenge, a maximum of about 6 months if sting challenge is performed right after reaching the maintenance dose
  A sensitization is considered predominant if the proportion of specific IgE to a single venom allergen is at least 65% of the specific IgE to the venom preparations.

SECONDARY OUTCOMES:
To evaluate if predominant sensitization to either Api m 1, Api m 2, Api m 3 or Api m 5 is a risk factor for treatment failure. | depends on the protocol used for VIT and the date of the sting challenge, a maximum of about 6 months if sting challenge is performed right after reaching the maintenance dose
To evaluate if low immunoglobulin G4 (IgG4) levels to bee venom or to Api m 1, Api m 2, Api m 3, Api m 5, or Api m 10 after VIT is a risk factor for treatment failure. | depends on the protocol used for VIT and the date of the sting challenge, a maximum of about 6 months if sting challenge is performed right after reaching the maintenance dose
To evaluate if systemic side effects are a risk factor for treatment failure. | depends on the protocol used for VIT and the date of the sting challenge, a maximum of about 6 months if sting challenge is performed right after reaching the maintenance dose
To evaluate if antihypertensive medication is a risk factor for treatment failure. | depends on the protocol used for VIT and the date of the sting challenge, a maximum of about 6 months if sting challenge is performed right after reaching the maintenance dose

CONTACTS AND LOCATIONS:
Locations (3):
- Department of Dermatology and Venerology, Medical University of Graz, Graz, Austria
- Elbe Klinikum Buxtehude, Buxtehude, Germany
- Hospital Universitario de Castellón, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Undecided